CLINICAL TRIAL: NCT05709600
Title: Dietary Interventions During Living Kidney Donations (DILKID Trial)
Brief Title: Dietary Interventions During Living Kidney Donations
Acronym: DILKID
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Roman Müller, Principal Investigator, University of Cologne
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V1.1-25052022
Record Dates: First submitted 2023-01-10; First posted 2023-02-02 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Living-Kidney Donors
Keywords: Transplant; Acute Kidney Injury; Kidney Dietary Interventions
MeSH Terms: conditions — Acute Kidney Injury | interventions — Diet, Ketogenic; Control Groups; Diet, Fat-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Fasting mimicking diet (Active Comparator): Human fasting mimicking diet (Prolon®) for five days prior to living kidney donation in donor: Day 1 of Prolon® supplies ~4600 kJ, day 2-5 provide ~3000kJ.
  Interventions: Dietary Supplement: Fasting mimicking diet
- Ketogenic diet (Active Comparator): Isocaloric, ketogenic diet 7 days prior to living kidney donation in the kidney donor with below 5% of energy from carbohydrate (<20g/day), approximately 15% from protein (<100g/day) and 80% from fat (>125g/day) without changes in caloric supply calculated by the Mifflin-St.Jeor formula achieved by the KetoCal 4:1 formula diet (Nutricia Milupa GmbH, Erlangen, Germany).
  Interventions: Dietary Supplement: Ketogenic diet
- Dietary restriction of sulfur containing amino acids (Active Comparator): Isocaloric, dietary restriction of sulfur containing amino acids in the donor without changes in caloric supply calculated by the Mifflin-St.Jeor formula achieved by the X Met X Cys Maxamaid formula diet (Nutricia Milupa GmbH, Erlangen, Germany).
  Interventions: Dietary Supplement: Dietary restriction of sulfur containing amino acids
- Control-Group (Active Comparator): Healthy, low-fat, moderate protein and high carbohydrate diet in the donor as described in the current nutritional recommendations of the American Diabetes Association achieved by the Fortimel® diet (Nutricia Milupa GmbH, Erlangen, Germany)
  Interventions: Dietary Supplement: Control Group ( healthy, low-fat, moderate protein and high carbohydrate diet)

INTERVENTIONS:
Dietary Supplement: Fasting mimicking diet — Intermittent fasting with human fasting mimicking diet (Prolon®) will be performed for five days prior to living kidney donation in the donor. Prolon® a plant-based diet designed to attain fasting-like effects while provide providing both macro- and micronutrient. Each participant will obtain Prolon® diet during the first visit and the diet will stored at the participant's home at room temperature. Additionally, the participant will receive a food plan for the exact consumption of the diet. Regular phone with a predefined standardized questionnaire will be used to determine each participant's well-being, as well as his or her dietary adherence. Furthermore, the participants will be asked to write down each consumed food items they are consuming in diet-book, which is handed to them during the first visit.
  The participants are only allowed to consume water, coffee or tea without sugar simultaneously to the Prolon® diet.
  Arms: Fasting mimicking diet
Dietary Supplement: Ketogenic diet — Isocaloric, ketogenic diet will be performed for seven days prior to living kidney donation in the donor.
  The ketogenic diet is based on the KetoCal 4:1 formula diet (Nutricia Milupa GmbH, Erlangen, Germany). Main fat sources are plant oils including palm oil and sunflower oils. The formula diet is provided as a powder that has to be mixed with water before use. To avoid a shortage in protein uptake supplement formula diets K-AM and Fortimel® (both Nutricia Milupa GmbH, Erlangen, Germany) will be used additionally. Salt uptake will be standardized employing either broths or salt tablets to not interfere with the steady-state salt and water homeostasis. A salt ingestion of 5g/day, which is common for western diets, is aimed at. The participants will receive a daily food plan by the dietetics at the University Hospital of Cologne to ensure standardized food consumption
  Arms: Ketogenic diet
Dietary Supplement: Dietary restriction of sulfur containing amino acids — Isocaloric, dietary restriction of sulfur containing amino acids will be performed for seven days prior to living kidney donation in the donor.
  A dietary restriction of sulfur containing amino acids without restriction in protein uptake will be achieved by following the X Met X Cys Maxamaid formula diet (Nutricia Milupa GmbH, Erlangen, Germany). The formula diet is provided as a powder that has to be mixed with water before use. A minimum of methionine and cysteine uptake (10% of the common uptake per day) will be achieved by consuming individuial calculated amounts of the Fortimel® formula diet (Nutricia Milupa GmbH, Erlangen, Germany). To avoid a restriction in fat and energy uptake additionally the Calogen and Duocal formula diets (both Nutricia Milupa GmbH, Erlangen, Germany) will be used. A salt ingestion of 5g/day, which is common for western diets, is aimed at. The participants will receive a daily food plan to ensure standardized food consumption.
  Arms: Dietary restriction of sulfur containing amino acids
Dietary Supplement: Control Group ( healthy, low-fat, moderate protein and high carbohydrate diet) — Participants in the control group will be instructed to adhere to a healthy, low-fat, moderate protein and high carbohydrate diet as described in current nutritional recommendations. The control diet will be based on the formula diet Fortimel® (Nutricia Milupa GmbH, Erlangen, Germany). Salt uptake will be standardized employing either broths or salt tablets to not interfere with the steady-state salt and water homeostasis. A salt ingestion of 5g/day, which is common for western diets, is aimed at.
  Arms: Control-Group

SUMMARY:
Monocentre, non-randomized, non-blinded, open-label interventional study to identification of relevant changes in molecular biology in proteome, phosphoproteome, lipidome, epigenome and transcriptome in pretransplant kidney biopsy samples in patients preconditioned by different dietary regimes (fasting mimicking diet vs. ketogenic diet vs. dietary restriction of sulfur containing amino acids vs. control patients)

DETAILED DESCRIPTION:
Acute kidney injury (AKI) is one of the most common disorders in hospitalized patients and the incidence of AKI is rapidly rising, especially among high-risk patients. In a meta-analysis including 49 million patients, AKI occurred in every fifth adult and in every third children suffering from an acute illness, defined as critical care with admission to the intensive care unit (ICU), cardiac surgery, trauma, heart failure or underlying disease within the field of haematology/oncology. AKI is associated with substantial mortality, even in non-ICU patients mortality ranges high between 10-20% and AKI severity is related to increased mortality. In addition, non-recovery of kidney function rates between 13-29% and progression to chronic kidney disease (CKD) requiring dialysis after AKI is common. Despite the considerable burden associated with AKI, effective therapeutic approaches, including prevention strategies, are currently lacking.

Since impaired cellular stress resistance contributes to AKI, preconditioning protocols that augment stress resistance such as caloric restriction (CR) are attractive strategies in the search for organprotection. CR protects from kidney damage in rodent models of AKI, induced by either ischemia-reperfusion injury or by injection of nephrotoxic cisplatin. However, the translation of this potential to the clinical setting has been hampered by both the limited understanding of the underlying mechanisms paired with the risk of malnourishment and significant comorbidity in the target patient population in terms of frailty, multi-morbidity or preoperative settings.

Based on more recent results regarding novel dietary regimens, three well-established targeted diets (a fasting mimicking diet, a ketogenic diet and the dietary restriction of sulfur-containing amino acids and the dietary restriction of branched chained amino acids), which already proved their safety and feasibility in both phase-II and I clinical trials, are promising novel targeted dietary strategies beyond CR.

Intermittent fasting with fasting mimicking diets enables the activation of cellular signal transduction similar to CR with high nourishment. Fasting mimicking diet efficiently protects from acute kidney injury in rodents. Human FMD (Prolon®) is a plant-derived diet to achieve fasting-like effects on serum levels of insulin growth factor-1 (IGF-1), insulin growth factor protein-1 (IGFP-1), glucose and ketone bodies, while providing both macro- und micronutrients. Intermitted fasting with fasting mimicking diets have extensively been studied in rodents. Additionally, phase-II and phase-I studies proofed safety, feasibility and favorable outcome in healthy volunteers and patients with autoimmune disorders or diabetes.

Ketogenic diets are high in fat and very low in carbohydrates and result in ketogenesis with the synthesis of ketone bodies, exceeding β-oxidation of fatty acids and anti-inflammation. Furthermore, ketogenic diets extend the lifespan in rodents with preserved physiological functions. Ketone bodies, such as β-hydroxybutyrate, suppress oxidative stress resulting in nephroprotection. Due to their additional neuroprotective effects, ketogenic diets have been in medical use in pharmacoresistant epilepsy proofing their feasibility and safety in humans. Moreover, ketogenic diets in women with ovarian and endometrial cancer revealed favorable effects on physical activity, perceived energy and food cravings. Considering that CR actually does induce ketogenesis due to feeding cycles, ketogenic diets are a key strategy that needs to be examined as a replacement for caloric restriction.

The amino acid methionine is the start codon in protein translation and is essential in the synthesis of the amino acid cysteine, which is also a precursor for glutathione and s adenosylmethionine, both needed in detoxification and methylation. Dietary restriction of these two sulfur-containing amino acids has been shown to be required for the beneficial effects of caloric restriction in a rodent model of liver damage. In addition, restriction in sulfur containing amino acids efficiently protects from acute kidney injury in rodents. Cysteine/methionine restriction activates the transsulfuration pathway resulting in the generation of hydrogen sulfide (H2S) and is associated with anti-inflammation, increased stress resistance, reduction of reactive oxygen species and alteration in lipid-metabolism. Sulfur containing amino acids are abundant in animal-derived protein, but also exist in certain vegetables, fruits and grains. A dietary restriction of sulfur containing amino acids can be achieved by a vegan-based diet without fish, meat, dairy products and certain plant-based foods as well as using specific formula diets Objective of the proof-of-principle, pilot-DILKID-trial is to decipher the underlying mediating mechanisms of different, well-established, dietary regimens as well as to prove their feasibility, tolerability and safety in nephrology patients. Additionally, the organprotective effects of those preoperative dietary interventions in terms of the transplant function in the kidney recipient will be analyzed. Inter-group differences on transcriptome, lipidome, metabolome, epigenome and (phospho-) proteome in the collected tissue (kidney, vessel and fat tissue), as well as in blood cells, plasma and serum will be compared between the different study arms.

In addition, the DILKID-trial aims to prove nephroprotective effects observed in rodent studies in humans and to correlate them with clinical surrogate parameters for kidney function. Another goal of our study consists in the identification of distinct metabolic pathways that are mediated by the dietary preconditioning strategies mentioned above and resulting in novel therapeutic approach protecting from AKI in nephrology patients

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years of age
* Planed living kidney transplantation (both donor and recipient are eligible)
* Written informed consent

Exclusion Criteria:

* Vegetarian lifestyle
* Body-Mass-Index (BMI) < 18.5 kg/m2
* Calorie-reduced diet within the preceding four weeks
* Underlying wasting syndrome
* Contraindication for enteral nutrition
* Known allergy to or intolerance of the ingredients of the diet used
* Pregnancy
* Breastfeeding
* Absence of safe contraceptive measures or non-occurrence of menopause (in women)
* Participation in other interventional trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Changes in proteome levels in pretransplant kidney biopsy samples | at baseline, at end of trial on day 9
  Measurement of proteome levels before and after the diet by mass spectrometry
Changes in phosphoproteome levels in pretransplant kidney biopsy samples | at baseline, at end of trial on day 9
  Measurement of phosphoproteome levels before and after the diet by mass spectrometry
Changes in lipidome levels in pretransplant kidney biopsy samples | at baseline, at end of trial on day 9
  Measurement of lipide levels before and after the diet by mass spectrometry
Changes in epigenome levels in pretransplant kidney biopsy samples | at baseline, at end of trial on day 9
  Measurement of epigenome levels before and after the diet by sequencing techniques
Changes in transcriptome levels in pretransplant kidney biopsy samples | at baseline, at end of trial on day 9
  Measurement of transcriptome levels before and after the diet by sequencing techniques

SECONDARY OUTCOMES:
Changes of Insulin-Like Growth-Factor Binding Protein C | at baseline, at the end of trial on day 9
  Measurement of Insulin-Like Growth Factor Binding Protein C in urine samples
Changes of Tissue Inhibitor of Metalloproteinases | at baseline, at the end of trial on day 9
  Determination in urine as predictive marker for acute kidney injury
Changes in Cystatin C | at baseline, at the end of trial on day 9
  Determination in blood samples as predictive marker for acute kidney injury
occurrence of acute kidney injury | at the end of trial on day 9
  Occurrence of acute kidney injury according to the Kidney Disease Improving Global Outcome (KDIGO) criteria
maximum serum creatinine in the recipient during hospitalization | during hospitalization, an average of 7 days, six weeks after transplantation and six month after transplantation
  Measurement of serum creatinine levels in blood samples
Feasibility of dietary interventions in every-day life | during 7 days of dietary intervention, at the end of trial on day 9
  Patient-reported feasibility will be measured using visual analogue scale (VAS), where min. 0 the worst outcome and max. 100 the best outcome means

CONTACTS AND LOCATIONS:
Overall Officials: Roman-Ulrich Müller, Prof. MD, Principal Investigator — Department II of Internal Medicine, University Hospital of Cologne
Locations (1):
- Department II of Internal Medicine, Center for Molecular Medicine Cologne (CMMC), University Hospital of Cologne, Cologne, Germany

IPD SHARING:
Plan to Share IPD: No